CLINICAL TRIAL: NCT02845258
Title: Treatment of Pancreatic Pseudocysts by Endoscopic Ultrasound-guided Drainage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Per Hedenström, MD, Sahlgrenska University Hospital
Other Study IDs: Dnr 573-09
Record Dates: First submitted 2016-07-20; First posted 2016-07-27 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Pancreatic Pseudocyst; Drainage
MeSH Terms: conditions — Pancreatic Pseudocyst | interventions — Self Expandable Metallic Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pancreatic pseudocyst fluid aspirate for culture and biochemical analysis. No DNA analysis.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Pancreatic pseudocyst drainage with a plastic or self-expandable metallic stent (SEMS) — Pancreatic pseudocyst drainage with a plastic or self-expandable metallic stent (SEMS):
  This procedure is to be regarded as a clinical routine procedure since a couple of years back. The type of stent (material? length? thickness?), the cyst appearance (large? infected? cyst wall thickness?) and the type of access (transgastric? transduodenal?) may however vary from patient to patient.
  In this study we perform EUS-drainage using different types of equipment on a wide range of pancreatic pseudocysts of different appearance and character. All procedures are performed as recommended. The very aim of the study is to investigate which technique and Equipment is to be preferred in different scenarios.

SUMMARY:
Patients may evolve pseudocysts of the pancreas secondary to a severe pancreatitis. In case of a symptomatic or infected pseudocyst, a therapeutic drainage of the cyst is indicated. In modern medicine the preferred way to perform such a drainage is by the means of endoscopic ultrasound (EUS). It is not precisely elucidated how this EUS-procedure should be performed in different scenarios. The cyst appearance and the drainage stents and/or technique may impact the clinical outcome.

This study is a prospective, single-center observational study on the outcome after EUS-guided drainage of pancreatic pseudocysts.

DETAILED DESCRIPTION:
Patintes referred to Sahlgrenska University hospital for an EUS-guided drainage of a pseudocyst are eligible for inclusion. The drainage is performed at the discretion of an experienced endosonographer. Thus, the equipment and the technique used may vary among patients but no randomization is done before the procedure. Intraprocedural variables are registered as well as data and outcome parameters from the clinical follow up according to below.

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years referred to the Sahlgrenska University hospital for the performance of an EUS-guided pancreatic pseudocyst drainage

Exclusion Criteria:

* Patients unwilling to participate or unable to understand or sign the informed consent
* Patients with no need for pseudocyst drainage as assessed by the endosonographer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients >18 years referred to the Sahlgrenska University hospital for the performance of an EUS-guided pancreatic pseudocyst drainage
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2006-01; Primary Completion 2021-10 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Short time complication rate | Uo to 48 hours
  The number of EUS-procedure-related complications such as bleeding, infection and death.
Repeated drainage frequency | Up to 3 months
  A successful drainage means no need for additional drainage procedures. The need for a repeated drainage is to be regarded as a therapeutic failure. The number of repeated procedures due to the need for additional drainage is recorded.

SECONDARY OUTCOMES:
Hospital stay | Up to 30 days
  The number of days spent in hospital post-EUS-drainage
Long time complication rate | Up to 6 months
  Infections and other complications related to the non-complete drainage of the pseudocyst after discharge from the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Riadh Sadik, Ass Prof, Study Director — Sahlgrenska University Hospital, Gothenburg
Locations (1):
- Endoscopy Department GEA, Sahlgrenska university Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No